CLINICAL TRIAL: NCT02253108
Title: Randomized Comparison of the Biolimus-eluting Biomatrix Neoflex™ og Everolimus-eluting SYNERGY™ Stents in All-comer Patients With Ischemic Heart Disease - The OCT SORT-OUT VIII
Brief Title: The OCT SORT-OUT VIII Study
Acronym: OCT SORT-OUT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Biosensors International (Other); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, MD, phd, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-125-14
Record Dates: First submitted 2014-09-09; First posted 2014-10-01 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Myocardial Infarction
Keywords: DES; Angina pectoris; Stent; Optical coherence tomography; Stent thrombosis
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SYNERGY drug eluting stent (Experimental): Everolimus eluting bioresorbable polymer stent
  Interventions: Device: Everolimus eluting bioresorbable polymer stent
- Biomatrix NeoFlex drug eluting stent (Experimental): Biolimus eluting bioresorbable polymer stent
  Interventions: Device: Biolimus eluting bioresorbable polymer stent

INTERVENTIONS:
Device: Everolimus eluting bioresorbable polymer stent
  Other Names: SYNERGY
  Arms: SYNERGY drug eluting stent
Device: Biolimus eluting bioresorbable polymer stent
  Other Names: Biomatrix NeoFlex
  Arms: Biomatrix NeoFlex drug eluting stent

SUMMARY:
The purpose of this study is to compare early vessel healing after implantation of SYNERGY drug eluting stent (DES) or BioMatrix NeoFlex DES at one and three months in two cohorts.

DETAILED DESCRIPTION:
Prospective, open label, single blind, randomized study with inclusion of 160 patients in two equal sized cohorts (A and B). Angiographic follow-up with optical coherence tomography (OCT) is performed at 1 month (Cohort A) and 3 months (Cohort B). Randomization 1:1 to SYNERGY or BioMatrix Neoflex. The Cohorts are included consecutively, Cohort A first.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years to be treated with one or more drug-eluting stents in a coronary artery at Aarhus University Hospital or Odense University Hospital

Exclusion Criteria:

* Age <18 years
* Do not wish to participate
* Unable to provide written informed consent
* Domicile outside Denmark
* Do not speak Danish
* Inclusion in the SORT-OUT VIII study
* Inclusion in other stent studies
* Expected survival <1 year
* Allergy to aspirin, clopidogrel, prasugrel or ticagrelor
* Hypersensitivity to everolimus or biolimus
* The operator wishes to use other DES
* Reduced renal function; creatinine> 120 mmol / L
* Only bare metal stent (BMS) implantation
* Only plain old balloon angioplasty (POBA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Coronary Stent Healing Index | 1 or 3 months
  Combined endpoint of vessel wall healing parameters assessed by optical coherence tomography (OCT)
Uncovered stent struts | 1 or 3 months
  Uncovered stent struts 2%=1, 5%=2, 10%=3, 15%=4, 20%=5, 25%=6, 30%=7, 35%=8, 40%=9
Uncovered stent struts in front of SBs, on acquired or persistent malapposed struts | 1 and 3 months
  Uncovered stent struts in front of side branchs (SB), on acquired or persistent malapposed struts10%=1, 20%=2, 30%=3 etc to 100%=0
Persistent malapposition | 1 and 3 months
  Persistent malapposition: >2 adjacent struts of at least 1 mm length =1; >2 mm=2; >3 mm=3
Neointimal thickness in one frame or lumen mean diameter stenosis | 1 and 3 months
  Neointimal thickness in one frame or lumen mean diameter stenosis >200=1; >300=2; >400=3 or diameter stenosis >50%=4; >75%=5
Acquired malapposition | 1 and 3 months
  Acquired malapposition: >2 adjacent struts of at least 1 mm length =2; > 2 mm=4; > 3 mm=6
Cumulated extra stent lumen increase in matched cross sectional analysis | 1 and 3 months
  Cumulated extra stent lumen increase in matched cross sectional analysis (measurement mean area)

SECONDARY OUTCOMES:
Malapposition | Baseline, 1 and 3 months
  Detectable separation between the vessel wall and strut in a cross section.
Coverage | Baseline, 1 and 3 months
  Detectable tissue covering the strut
Fracture | Baseline, 1 and 3 months
  Discontinuity of a strut evaluated by 3D reconstruction
Neointimal thickness (NIT) | Baseline, 1 and 3 months
  Thickness of intima from leading strut surface to lumen boarder
Lumen area | Baseline, 1 and 3 months
  Area of lumen in cross section
Stent area | Baseline, 1 and 3 months
  Area of stent in cross section
Area stenosis (AS) % | Baseline, 1 and 3 months
  Minimal luminal area/reference area (interpolated)
Minimum expansion of the stent | Baseline, 1 and 3 months
  Expressed as absolute area and percentage of the closest reference area
Late recoil | Baseline, 1 and 3 months
  Loss in stent area from baseline to follow-up
Lumen late loss | Baseline, 1 and 3 months
  Loss in minimal lumen area from baseline to follow-up
Extra stent lumen | Baseline, 1 and 3 months
  Area outside stent boarder limited by lumen boarder
Evaginations | Baseline, 1 and 3 months
  Counts and descriptive by size (volume and depth)
Thrombus on struts | Baseline, 1 and 3 months
  In final OCT after implantation and at follow-up
Acute expansion and late recoil | Baseline, 1 and 3 months
  In segments with; 1)calcified plaque, 2)lipid plaque, 3)area after predilatation <30% of reference area, 4)stenosed segments (>50% AS) with no dissections after predilatation
Target Lesion Failure (TLF) | Within 12 months
  Stent related combined endpoint of Target Lesion Failure (TLF) hierarchically as cardiac death, non-index procedure related AMI (defined as AMI not clearly related to another lesion than the target lesion), or Target Lesion Revascularisation (TLR) (by PCI or CABG - TLR if significant stenosis + 5mm distal/proximal)
Cardiac death | Baseline, 12, 24, 36, 48 and 60 months
  Stent related, major adverse cardiac events (MACE), serious complication at procedure
Non-index procedure related acute myocardial infarction (AMI) | Baseline and within 12, 24, 36, 48 and 60 months
  Defined as AMI not clearly related to another lesion than the target lesion
Target Lesion Revascularisation (TLR) | Baseline and within 12, 24, 36, 48 and 60 months
  New revascularisation of TLR by percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) (TLR if significant stenosis += 5 mm distal/proximal)
All-cause death | 12, 24, 36, 48 and 60 months
Stent thrombosis | Baseline, 1, 12, 24, 36, 48 and 60 months
  According to ARC criteria
Device success rate | Baseline
  Defined as the frequency of successful implantation with residual stenosis <20% of the study stent in all the stenoses scheduled to be treated
Procedural success rate | Baseline
  Defined as the frequency of successful implantation with residual stenosis <20% of the study stent in all the stenoses scheduled to be treated and without serious complications

CONTACTS AND LOCATIONS:
Overall Officials: Evald H Christiansen, MD, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Skejby, Aarhus
  - Odense University Hospital, Odense